CLINICAL TRIAL: NCT00160160
Title: A Multi-Center, Double-Blind, Randomized Study Comparing the Efficacy of Combination Therapy of Eprosartan Respectively Ramipril With Low-Dose Hydrochlorothiazide and Moxonidine on Blood Pressure Levels in Patients With Hypertension and Associated Diabetes Mellitus Type 2
Brief Title: Comparison of Eprosartan/HCT Versus Enalapril/HCT in Hypertensives With Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S171.3.012; 2004-00703-18
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension; Type 2 Diabetes
Keywords: comparator trial; hypertension; diabetes; blood pressure
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Drug: eprosartan/HCTZ

SUMMARY:
This study is to demonstrate the superiority of combination of eprosartan/HCTZ versus ramipril/HCTZ.

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension,
* diabetes type 2

Exclusion Criteria:

* severe cardiovascular disease,
* grade 3 hypertension,
* secondary hypertension,
* abnormal liver enzymes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2004-10

PRIMARY OUTCOMES:
Blood pressure reduction

SECONDARY OUTCOMES:
Comparison of responder rates

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (63):
- Canada (6):
  - Site 26, Calgary
  - Site 27, Montreal
  - Site 30, Québec
  - Site 31, Thornhill
  - Site 28, Vancouver
  - Site 29, Winnipeg
- Denmark (3):
  - Site 39, Holbæk
  - Site 38, Roskilde
  - Site 40, Viborg
- France (15):
  - Site 4, Anzin
  - Site 3, Blois
  - Site 10, Chemellier
  - Site 11, Cholet
  - Site 15, Cholet
  - Site 16, Cholet
  - Site 14, La Jubaudière
  - Site 13, Le Mesnil-en-Vallée
  - Site 7, Mûrs-Erigné
  - Site 12, Saint Pierre Montlim
  - Site 9, Saumur
  - Site 8, Segré
  - Site 6, Thouars
  - Site 2, Tours
  - Site 5, Vieux-Condé
- Germany (9):
  - Site 20, Bad Muenster
  - Site 22, Flörsheim
  - Site 19, Kirweiler
  - Site 21, Lambrecht
  - Site 25, Lindau
  - Site 24, Lutherstadt
  - Site 18, Lüneburg
  - Site 17, Riesa
  - Site 23, Waldbrunn
- Italy (7):
  - Site 62, Bologna
  - Site 60, Napoli
  - Site 58, Padua
  - Site 59, Palermo
  - Site 63, Pavia
  - Site 61, Pisa
  - Site 64, Torino
- Norway (4):
  - Site 43, Ålesund
  - Site 42, Bergen
  - Site 44, Horten
  - Site 41, Skedsmokorset
- Spain (7):
  - Site 55, Badajoz
  - Site 51, Badalona
  - Site 56, Barcelona
  - Site 57, Barcelona
  - Site 54, Ciudad Real
  - Site 53, Granada
  - Site 52, Madrid
- Sweden (6):
  - Site 48, Ängelholm
  - Site 47, Gothenburg
  - Site 46, Helsingborg
  - Site 45, Kristianstat
  - Site 50, Malmo
  - Site 49, Stockholm
- United Kingdom (6):
  - Site 33, Aberdeen
  - Site 36, Bath
  - Site 37, Liverpool
  - Site 34, Manchester
  - Site 32, Oldham
  - Site 35, Rugby